CLINICAL TRIAL: NCT06241352
Title: A Prospective Clinical Trial of Statin Addition to Chemotherapy for Advanced Pancreatic Cancer
Brief Title: Statin Addition to Chemotherapy for Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Guo ShiWei, Associate Chief Doctor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChanghaiH-PP13
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Advanced Pancreatic Cancer
Keywords: advanced pancreatic cancer; statin; chemotherapy resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Statin addition to chemotherapy (Experimental): Chemotherapy plus atorvastatin was used in locally advanced pancreatic cancer.
  Interventions: Drug: statin addition to chemotherapy

INTERVENTIONS:
Drug: statin addition to chemotherapy — Chemotherapy was administered along with 80mg of atorvastatin per day. Atorvastatin was discontinued when CA19-9 levels (with CA19-9 negative patients referenced against CEA or CA-125) rose more than 20% above baseline.

SUMMARY:
The results of previous studies conducted by our team have revealed that the use of statins can more effectively hinder the growth of drug-resistant pancreatic cancer cells. The primary objective of this study was to investigate the role of statins in treating pancreatic cancer by assessing the safety and therapeutic impact of combining chemotherapy with statins in patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
The poor prognosis of pancreatic cancer is not just because of the high malignancy of the tumor itself, but also its poor response to chemotherapy. Gemcitabine and fluorouracil are the primary drugs utilized in pancreatic cancer treatment, and combination chemotherapy predominantly revolves around these two drugs. Nevertheless, findings from clinical studies reveal that approximately one-third of pancreatic cancer patients display resistance to chemotherapy, with the majority of the remaining patients eventually developing secondary resistance within six months following treatment. Consequently, chemotherapy resistance constitutes a significant factor contributing to the poor prognosis of pancreatic cancer patients.

Our research team established a biobank containing over 300 pancreatic cancer organoids. Using high-throughput drug sensitivity detection techniques, the investigators assessed the sensitivity of 177 pancreatic cancer organoids to five commonly used chemotherapeutics and 84 tumor-related drugs or regimens. The findings suggest that pancreatic cancer organoids that are generally resistant to chemotherapy drugs exhibit sensitivity to statins. These findings indicate that combining chemotherapy with statins may enhance the therapeutic effect for pancreatic cancer patients. Previous studies have also reported the potential therapeutic effects of statins in colorectal, lung and breast cancer.

In summary, chemotherapy resistance is a significant factor contributing to the poor prognosis of pancreatic cancer. Building on previous research conducted by our team, this study aims to investigate the role of statins in pancreatic cancer through a single-arm clinical trial, with the goal to investigate the role of statins in treating pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old and ≤80 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or
* Histologically or cytologically confirmed local advanced/metastatic pancreas adenocarcinoma.
* Imaging studies confirmed the diagnosis of locally advanced or metastatic pancreatic cancer patients.
* The patients were in the plateau stage after chemotherapy, as indicated by the CA19-9 values (with CA19-9 negative patients referenced against CEA or CA-125) fluctuating by less than 20% over an interval of more than 3 weeks.
* Life expectancy of greater than 90 days, as judged by the investigator.
* Routine blood test: absolute neutrophil count>1500/mm3, platelet>100000/ mm3.
* Normal liver function: serum total bilirubin≤2.0mg/dl, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <3 times of the upper limit of normal value.
* Normal kidney function: serum creatinine<1.5 times of the upper limit of normal value or creatinine clearance rate>45ml/min.
* No severe comorbidities.

Exclusion Criteria:

* Patients with poor condition can not tolerate chemotherapy.
* Patients who have previously taken lipid-lowering drugs (such as statins, fibrates, ezetimibe, or PCSK9 inhibitors).
* Patients who are taking warfarin, verapamil, clopidogrel, digoxin, amiodarone, etc.
* Impaired organ functions: heart failure (New York Heart Association III- IV), coronary heart disease, myocardial infarction within 6 months, severe cardiac arrhythmia and respiratory failure.
* Patients diagnosed with other cancer within 5 years.
* Patients who are pregnant or breastfeeding.
* Patients enrolled in other clinical trials or incompliant of regular follow up.
* Patients who did not provide an informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Decrease rate of CA19-9 (with CA19-9 negative patients referenced against CEA or CA-125) | 1-2 month
  The proportion of patients with a decrease of over 20% in CA19-9 (with CA19-9 negative patients referenced against CEA or CA-125) one month after the start of treatment.

SECONDARY OUTCOMES:
Event-free Survival | 1 year
  Defined as the time between signing the informed consent form to the first documentation of event where events considered are 1) disease progression (local recurrence, new lesions or distant metastasis), 2) a second malignant tumor occurs, or 3) death due to any cause.
Overall survival | 2 years
  Defined as the time between signing the informed consent form and death due to various causes.
Disease control rate | 6 months
  Defined as the proportion of patients who achieved complete response (CR), partial response (PR) and stable disease (SD) according to RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Jin, MD, Principal Investigator — Changhai Hospital, Shanghai, China
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No